CLINICAL TRIAL: NCT03627650
Title: Fat Grafting in Immature Skin-grafted Burn Scars: a Randomised Controlled Clinical Trial
Brief Title: Fat Grafting in Skin-grafted Deep Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Phillip Blondeel, Clinical Professor, Head of Plastic Surgery, Principal Investigator, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 2010/ 572
Record Dates: First submitted 2017-10-06; First posted 2018-08-13 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Burn Scar
Keywords: burn; scar; fat; grafting
MeSH Terms: conditions — Burns; Cicatrix; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: 2 skin zones per participant, A and B, 1 is treated, 1 is placebo coin toss determines which zone will be treated, this information is kept in sealed envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 group of 15 patients (Experimental): procedure/surgery: fat grafting injection of scar
  Interventions: Procedure: lipofilling/ fat grafting
- Same group of 15 patients (Experimental): procedure/surgery: placebo injection of scar
  Interventions: Procedure: placebo injection

INTERVENTIONS:
Procedure: lipofilling/ fat grafting — liposuction, processing/ cleaning of fat tissue; reinjection with sharp needle transcutaneous
  Arms: 1 group of 15 patients
Procedure: placebo injection
  Arms: Same group of 15 patients

SUMMARY:
fat grafting in human skin-grafted immature burn scars histological, clinical and photographic follow-up

DETAILED DESCRIPTION:
Objective: A randomised clinical trial was performed to determine the effect of autologous fat grafting on scar formation in early skin-grafted deep burn wounds.

Methods: Included patients received split-thickness skin grafting procedures for deep burn wounds less than 3 months ago. A homogenous scar area in each patient was divided into two equal parts. One part was treated with transcutaneous sharp needle autologous fat grafting, the adjacent part with transcutaneous saline injection as control. Results were evaluated by clinical assessment with scar scale questionnaires, histological examination, and objective scar assessment with Cutometer, Mexameter, Tewameter and Corneometer.

ELIGIBILITY:
Inclusion Criteria:

* early skin-grafted deep burn scars
* otherwise healthy

Exclusion Criteria:

* concomitant disease

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Improvement of scar quality by histological assessment | 6 months
  histology of scar tissue, scoring by 2 independent blinded anatomopathologists, (numerical scoring of fibroblast activity, collagen and elastin organisation, vascularity) scoring range min 1(close to normal tissue) - 3 (scar characteristics)
improvement of scar quality by physiological testing with cutometer | 6 months, 1 year
  measures elasticity of the scar; micrometer; higher values better outcome
Improvement of scar quality by subjective evaluation with numerical Vancouver Scar Scale | 1 year
  numerical score 0 to 13; ranges vascularity, height/thickness, pliability, and pigmentation
Improvement of scar quality by subjective evaluation with numerical POSAS (Patient and Observer Scar Assessment Scale) Scale | 1 year
  numerical score 5 to 50: VSS plus surface area; patient assessments of pain, itching, color, stiffness, thickness, relief
improvement of scar quality by physiological testing with TEWA-meter (Trans Epidermal Water Loss-meter) | 6 months, 1 year
  measures transepidermal water loss; g/m2/h; higher values worse outcome
physiological testing of scar tissue by corneometer | 6 months, 1 year
  measures hydration of the epidermis; corneometer units, higher values better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Maarten AJ Doornaert, MD, Principal Investigator — UGent University Hospital

IPD SHARING:
Plan to Share IPD: No